CLINICAL TRIAL: NCT02045537
Title: Retrospective Study to Determine the Incidence of Bone Fractures in HIV-infected Patients in Spain
Acronym: INFOHS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Other Study IDs: GESIDA-7312
Record Dates: First submitted 2014-01-15; First posted 2014-01-27 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: HIV
Keywords: HIV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fractures: Patients in follow up from 1st Jan 1997 to 1st Jan 2012 with any fracture (pathologic)

SUMMARY:
Study to determine the incidence of Bone Fractures in HIV infected patients in Spain

DETAILED DESCRIPTION:
Study to know the incidence of bone fractures in HIV patients, determine associate factors to bone fractures, the type of patients with fractures.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Signed ICF
* Patient that fulfill these:

  * Osteroporosis associated fracture
  * Enough information close to the moment of the fracture

Exclusion Criteria:

* patients with cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients HIV in followed up betwen 1 Jan 1997 and 1 Jan 2012
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-06; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
number of HIV patients with bone fractures | 18 years
  To know the incidence of bone fractures in HIV infected patients in Spain

SECONDARY OUTCOMES:
The number of fractures associated to determine factors | 18 years
  Determine associate factors to fractures
Number of patients with fractures | 18 years
  Determine the profile of patients with fractures

CONTACTS AND LOCATIONS:
Locations (24):
- Spain (24):
  - H. de Elche, Elche, Alicante
  - H. Marina Baixa, Villajoyosa, Alicante
  - H. Germans Trias i Pujol, Badalona, Barcelona
  - H. de Mataró, Mataró, Barcelona
  - H. Sabadell, Sabadell, Barcelona
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, La Coruña
  - H. Clinico Universitario Santiago de Compostela, Santiago de Compostela, La Coruña
  - H. Principe de Asturias, Alcalá de Henares, Madrid
  - H. Fundación de Alcorcón, Alcorcón, Madrid
  - H. Severo Ochoa, Leganés, Madrid
  - H. Clinic i Provincial, Barcelona
  - H. Santa Creu i Sant Pau, Barcelona
  - H. Virgen de la Luz, Cuenca
  - H. San Pedro de Logroño, Logroño
  - H. Clinico San Carlos, Madrid
  - H. Universitario Clínico San Carlos, Madrid
  - H. Universitario Infanta Leonor, Madrid
  - H. Universitario La Paz, Madrid
  - H. Arnau de Vilanova, Valencia
  - H. Clinico de Valencia, Valencia
  - H. La Fe, Valencia
  - H. Rio Hortega, Valladolid
  - H. Universitario Araba, Vitoria-Gasteiz
  - H. Lozano Blesa, Zaragoza